CLINICAL TRIAL: NCT05247125
Title: The Role of Circadian Factors in Regulation of Neuroplasticity in Ischemic Stroke (Interventional)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Lyudmila Korostovtseva, Senior Researcher, Department for Hypertension, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-75-10173-1 (interventional)
Record Dates: First submitted 2022-01-26; First posted 2022-02-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke, Acute; Sleep Disorders, Circadian Rhythm
Keywords: circadian misalignment; neuroplasticity; melatonin; light therapy; circadian disorder
MeSH Terms: conditions — Ischemic Stroke; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: patients will be randomized into 4 parallel groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Blue light exposure + Melatonin treatment (Experimental): The participants will receive the combination of blue light exposure according to the protocol described by Killgore et al. (2020) and 3 mg of melatonin 1 hour before going to sleep (approximately at 20:00) (Ramos et al 2020) for 14 days
  Interventions: Combination Product: Blue light exposure + Melatonin treatment
- Melatonin treatment (Experimental): The participants will receive 3 mg of melatonin 1 hour before going to sleep (approximately at 20:00) (Ramos et al 2020) and the morning placebo-light exposure according to the protocol described by Killgore et al. (2020) for 14 days
  Interventions: Drug: Melatonin treatment
- Blue light exposure (Experimental): The participants will receive the morning blue light exposure according to the protocol described by Killgore et al. (2020) for 14 days and placebo pill 1 hour before going to sleep (approximately at 20:00)
  Interventions: Device: Blue light exposure
- Placebo group (Placebo Comparator): The participants will receive placebo light exposure in the morning (lamp turned off) and placebo pill treatment in the evening for 14 days
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Blue light exposure + Melatonin treatment — 3 mg Melatonin pill will be given 1 hour before going to bed. Blue light exposure will be performed during 30-minute sessions with the use of the lamps (Lumie/Vitamin L) in the morning.
  Arms: Blue light exposure + Melatonin treatment
Drug: Melatonin treatment — 3 mg Melatonin pill will be given 1 hour before going to bed.
  Other Names: Melaxen
  Arms: Melatonin treatment
Device: Blue light exposure — Blue light exposure will be performed during 30-minute sessions with the use of the lamps (Lumie/Vitamin L) in the morning.
  Other Names: Lamps Lumie/Vitamin L
  Arms: Blue light exposure
Combination Product: Placebo — Placebo light exposure will be performed by using lamp turned off; and placebo pill will be given in the evening
  Arms: Placebo group

SUMMARY:
There is a lack of complex studies which could establish the association between genetic circadian factors with the features and short-term outcomes of ischemic stroke, as well as the effects of various auxiliary therapies for circadian rhythm modulation for neuroplasticity enhancement and improvement of short-term outcomes in ischemic stroke.

The main research hypothesis is that circadian factors influence the recovery from ischemic stroke via sleep-mediated regulation of synaptic plasticity.

The project aims at the investigation of the influence of combined melatonin therapy and blue light exposure on molecular circadian biomarkers, sleep characteristics, neuroplasticity markers and stroke outcome in acute stroke patients.

This study is a prospective, interventional, randomized placebo-controlled trial.

DETAILED DESCRIPTION:
The study will investigate the influence of combined blue light exposure and melatonin therapy on molecular biomarkers of circadian rhythms, sleep characteristics and stroke outcome in acute stroke patients This study is designed as a prospective study in acute stroke patients (approx 80 patients) admitted to the Stroke Unit. After initial assessment, the participants will be randomly assigned in 4 groups (the treatment or control) with approx.20 participants in each group.

In all participants, the following parameters will be assessed: medical records, stroke characteristics, sleep characteristics, cardiovascular circadian rhythms and blood samples for the evaluation of circadian molecular biomarkers at baseline and 14 days after inclusion. Stroke outcomes will be reassessed at 3-month follow-up.

The following associations will be assessed:

* the role of blue light exposure and melatonin treatment for stroke outcome
* the role of blue light exposure and melatonin treatment in the modulation of sleep parameters in acute stroke
* the association of molecular biomarkers of circadian rhythms with stroke outcome (the difference in neurological and functional deficit from admission to 14 and 90 days after study inclusion), with stroke characteristics (stroke subtype and neuroimaging stroke parameters, routine protocol) and with sleep characteristics.
* the association of sleep characteristics with stroke outcome (the difference in neurological and functional deficit from admission to 14 and 90 days after stroke) and with stroke characteristics (stroke subtype and neuroimaging stroke parameters, routine protocol).

ELIGIBILITY:
Inclusion Criteria:

* acute (symptom onset to admission <1 days) ischemic stroke
* ischemic stroke affecting the branches of anterior cerebral artery, middle cerebral artery and posterior cerebral artery
* age 18-80 years
* moderate or severe stroke (National Institutes of Health Stroke Scale, NIHSS>=5)
* intravascular stroke treatment with thrombolysis or thrombectomy leading to satisfactory reperfusion (if applicable)
* informed consent

Exclusion Criteria:

* secondary parenchymal hemorrhage (>hemorrhage index (HI)-2)
* clinically unstable or life-threatening conditions
* previous stroke in the last 6 months
* known progressive neurological diseases
* known psychiatric diseases
* concomitant benzodiazepine medication
* drug or alcohol abuse
* pregnancy
* inability to participate in the study
* severe sensory aphasia
* melatonin intake at/before admission
* light therapy use at/before admission
* blindness
* severe sleep-disordered breathing (apnea-hypopnea index >=30/h)
* contraindications to light therapy (severe retinopathy, epilepsy, porphyria, intake of drugs with photosensitizing effects)
* contraindications to melatonin intake (severe bronchial asthma, severe autoimmune disorders, chronic kidney disease 3b stage and higher, leukosis)
* congestive heart failure with reduced ejection fraction (<=45%) or New York Heart Association (NYHA) classification III-IV functional class.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the value of National Institutes of Health Stroke Scale from baseline to 14 days after inclusion | From baseline to 14 days after treatment initiation
  National Institutes of Health Stroke Scale (NIHSS) is a tool used to objectively quantify the impairment caused by a stroke, 0-42 scores, higher scores characterize worse impairment
Stroke-related disability assessed by the change in modified Rankin scale from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  values of modified Rankin scale (scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke, from 0 (no symptoms) to 6 (dead) points)
Stroke-related disability assessed by the change in Rivermead Mobility Index from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Rivermead Mobility Index (a standardized scale used to assess mobility in patients with neurological deficits, a maximum of 15 points is possible; higher scores indicate better mobility performance)
Stroke-related disability assessed by the change in Barthel Index from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Barthel Index (a common scale used to measure performance in activities of daily living, 0-100 scores, higher scores define better performance)

SECONDARY OUTCOMES:
Change in Psychomotor vigilance task (mean reaction time) from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  The psychomotor vigilance task is a sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus, the outcome (mean reaction time) is measured in msec
Change in Psychomotor vigilance task (mean reaction time) from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  The psychomotor vigilance task is a sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus, the outcome (mean reaction time) is measured in msec
Change in Kraepelin test from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Kraepelin test is the test in which the examinee performs a simple single-digit addition. The outcome is the number of correct and incorrect addition operations per each 30 sec and during the whole task, performance index (number of correct addition operations during second part of task / number of correct addition operations during first part of task)
Change in Kraepelin test from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Kraepelin test is the test in which the examinee performs a simple single-digit addition. The outcome is the number of correct and incorrect addition operations per each 30 sec and during the whole task, performance index (number of correct addition operations during second part of task / number of correct addition operations during first part of task)
Change in Trail Making test from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Trails Making Test (Trails) is a neuropsychological test of visual attention and task switching. It can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning
Change in Trail Making test from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Trails Making Test (Trails) is a neuropsychological test of visual attention and task switching. It can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. Execution time will be assessed (in msec)
Change in Victoria Stroop test from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Victoria Stroop is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference. Execution time will be measured. (in msec)
Change in Victoria Stroop test from baseline to 90 days after inclusion | From baseline to 90±7 day after inclusion
  Victoria Stroop is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference. Execution time will be measured. (in msec)
Change in Hopkins Verbal Learning Test (Revised) from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Hopkins Verbal Learning Test - Revised brief assessment of immediate recall, delayed recall and delayed recognition. The number of words recalled will be assessed.
Change in Hopkins Verbal Learning Test (Revised) from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Hopkins Verbal Learning Test - Revised brief assessment of immediate recall, delayed recall and delayed recognition. The number of words recalled will be assessed.
Change in Brief Visuospatial Memory Test (Revised) from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Brief Visuospatial Memory Test (Revised)is a commonly used, commercialized, assessment tool to measure visuospatial learning and memory abilities across research and clinical settings. The number of figures will be assessed.
Change in Brief Visuospatial Memory Test (Revised) from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Brief Visuospatial Memory Test (Revised)is a commonly used, commercialized, assessment tool to measure visuospatial learning and memory abilities across research and clinical settings. The number of figures will be assessed.
Change in Wechsler Memory Scale (Revised) from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  Wechsler Memory Scale - Revised is a neuropsychological test designed to measure different memory functions in a person. A composite score will be assessed.
Change in Wechsler Memory Scale (Revised) from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Wechsler Memory Scale - Revised is a neuropsychological test designed to measure different memory functions in a person. A composite score will be assessed.
Change in Corsi block-tapping test from baseline to 14 days after treatment initiation | From baseline to 14 days after treatment initiation
  The Corsi block-tapping test is a psychological test that assesses visuo-spatial short term working memory. The visual span raw score will be assessed.
Change in Corsi block-tapping test from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  The Corsi block-tapping test is a psychological test that assesses visuo-spatial short term working memory. The visual span raw score will be assessed.
Change from baseline in objective sleep duration assessed by polysomnography | From baseline to 14 days after treatment initiation
  Sleep duration (minutes)
Change from baseline in objective sleep efficiency assessed by polysomnography | From baseline to 14 days after treatment initiation
  sleep efficiency (%)
Change from baseline in objective sleep latency assessed by polysomnography | From baseline to 14 days after treatment initiation
  sleep latency (minutes)
Change from baseline in sleep S1 stage duration assessed by polysomnography | From baseline to 14 days after treatment initiation
  S1 sleep stage percentage of total sleep time (%)
Change from baseline in sleep S2 stage duration assessed by polysomnography | From baseline to 14 days after treatment initiation
  S2 sleep stage percentage of total sleep time (%)
Change from baseline in sleep S3 stage duration assessed by polysomnography | From baseline to 14 days after treatment initiation
  S3 sleep stage percentage of total sleep time (%)
Change from baseline in rapid eye movement (REM) sleep stage duration assessed by polysomnography | From baseline to 14 days after treatment initiation
  Rapid eye movement (REM) sleep stage percentage of total sleep time (%)
Change from baseline in wake-after-sleep-onset time assessed by polysomnography | From baseline to 14 days after treatment initiation
  wake after sleep onset time (minutes)
Change from baseline in arousal index assessed by polysomnography | From baseline to 14 days after treatment initiation
  Arousal index (episodes/hour of sleep)
Change in emotional outcome assessed by Hospital anxiety and depression scale from baseline to 90 days after inclusion | from baseline to 14 days after treatment initiation
  Hospital anxiety and depression scale is used to determine the levels of anxiety and depression. It is a 14-item scale; Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression, higher scores indicate worse situation
Change in emotional outcome assessed by Hospital anxiety and depression scale from baseline to 14 days after treatment initiation | From baseline to 90±7 days after inclusion
  Hospital anxiety and depression scale is used to determine the levels of anxiety and depression. It is a 14-item scale; Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression, higher scores indicate worse situation
Assessment of mood by change in Visual Analogue Mood Scale from baseline to 14 days after treatment initiation | from baseline to 14 days after treatment initiation
  Visual Analogue Mood Scale is a reliable and valid measure of eight specific mood states: Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense. The score for each mood ranges from 0 to 100 (100 mm vertical line), with 100 representing a maximal level of that mood and zero representing a minimal level (or absence) of that mood
Assessment of mood by change in Visual Analogue Mood Scale from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Visual Analogue Mood Scale is a reliable and valid measure of eight specific mood states: Afraid, Confused, Sad, Angry, Energetic, Tired, Happy, and Tense. The score for each mood ranges from 0 to 100 (100 mm vertical line), with 100 representing a maximal level of that mood and zero representing a minimal level (or absence) of that mood
Change in the value of National Institutes of Health Stroke Scale from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  National Institutes of Health Stroke Scale (NIHSS) is a tool used to objectively quantify the impairment caused by a stroke, 0-42 scores, higher scores characterize worse impairment
Change in modified Rankin scale from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  values of modified Rankin scale (scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke, from 0 (no symptoms) to 6 (dead) points)
Change in Rivermead Mobility Index from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Rivermead Mobility Index (a standardized scale used to assess mobility in patients with neurological deficits, a maximum of 15 points is possible; higher scores indicate better mobility performance)
Change in Barthel Index from baseline to 90 days after inclusion | From baseline to 90±7 days after inclusion
  Barthel Index (a common scale used to measure performance in activities of daily living, 0-100 scores, higher scores define better performance)

OTHER OUTCOMES:
Change from baseline in time in bed assessed by actigraphy | from baseline to 14 days after treatment initiation
  time in bed (minutes)
Change from baseline in total sleep time assessed by actigraphy | from baseline to 14 days after treatment initiation
  total sleep time (minutes)
Change from baseline in sleep efficiency assessed by actigraphy | from baseline to 14 days after treatment initiation
  sleep efficiency (%)
Change from baseline in sleep onset latency assessed by actigraphy | from baseline to 14 days after treatment initiation
  sleep onset latency (min)
Change from baseline in number of awakenings assessed by actigraphy | from baseline to 14 days after treatment initiation
  number of awakenings
Change from baseline in mean motor activity assessed by actigraphy | from baseline to 14 days after treatment initiation
  mean motor activity (units)
Change from baseline in Sleep Quality Score assessed by questionnaire Pittsburgh Sleep Quality Index | from baseline to 14 days after treatment initiation
  Pittsburgh Sleep Quality Index is a self-rated questionnaire which assesses subjective sleep quality and disturbances over a 1-month time interval, Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score indicating worse sleep quality
Change from baseline in daytime sleepiness assessed by Epworth Sleepiness Scale | from baseline to 14 days after treatment initiation
  Epworth Sleepiness Scale is a common tool to assess sleepiness; 0-24 points, higher score indicate greater sleepiness
Change from baseline in fatigue severity assessed by Fatigue severity Scale | from baseline to 14 days after treatment initiation
  Fatigue severity Scale is a common 9-item tool used to determine and quantify fatigue as subjective feeling of exhaustion, persisting lack of energy and rapid inanition, 9-63 points, higher score indicates more severe fatigue
Change from baseline in Insomnia severity index | from baseline to 14 days after treatment initiation
  Insomnia severity index is a 7-item tool to assess the severity of insomnia, 0-5 points per each item, higher score indicates more severe insomnia
Change from baseline in sensorimotor assessment of upper limbs | from baseline to 14 days after treatment initiation
  Sensorimotor assessment of upper limbs by Fugl-Meyer is a stroke-specific, performance-based impairment index. The total possible scale score is 226
Change from baseline in melatonin curve secretion | from baseline to 14 days after treatment initiation
  salivary melatonin levels samples collected every 3 hours for 24 hours at study inclusion and at 14 days after study inclusion
Change from baseline in cortisol curve secretion | from baseline to 14 days after treatment initiation
  salivary cortisol sampled every 3 hours for 24 hours at study inclusion and at 14 days after study inclusion
Change from baseline in circadian brain-derived neurotrophic factor messenger ribonucleic acid (mRNA) expression | from baseline to 14 days after treatment initiation
  Brain-derived neurotrophic factor messenger ribonucleic acid (mRNA) expression will be measured in blood samples taken every 4 hours for 24 hours at study inclusion and at 14 days after study inclusion
Change from baseline in circadian clock gene CLOCK messenger ribonucleic acid (mRNA) expression | from baseline to 14 days after treatment initiation
  clock gene CLOCK messenger ribonucleic acid (mRNA) expression will be measured in blood samples taken every 4 hours for 24 hours at study inclusion and at 14 days after study inclusion
Change from baseline in circadian clock gene Bmal1 messenger ribonucleic acid (mRNA) expression | from baseline to 14 days after treatment initiation
  clock gene Bmal1 messenger ribonucleic acid (mRNA) expression will be measured in blood samples taken every 4 hours for 24 hours at study inclusion and at 14 days after study inclusion
Change from baseline in circadian Melatonin receptor messenger ribonucleic acid (mRNA) expression | from baseline to 14 days after treatment initiation
  Melatonin receptor messenger ribonucleic acid (mRNA) expression will be measured in blood samples taken every 4 hours for 24 hours at study inclusion and at 14 days after study inclusion
Change in psychophysiological state: heart rate variability assessed by biofeedback method from baseline to 14 days | from baseline to 14 days after treatment initiation
  heart rate variability assessed by electrocardiogram (maximum heart rate - minimum heart rate, beats per minute)
Change in psychophysiological state: heart rate variability assessed by biofeedback method from baseline to 90 days after inclusion | from baseline to 90±7 days after inclusion
  heart rate variability assessed by electrocardiogram (maximum heart rate - minimum heart rate, beats per minute)
Change in psychophysiological state: respiratory movement amplitude assessed by biofeedback method - from baseline to 14 days | from baseline to 90±7 days after treatment initiation
  respiratory movement amplitude assessed by respiratory rate abdominal and thoracic sensors (units)
Change in psychophysiological state: respiratory movement amplitude assessed by biofeedback method- from baseline to 90 days | from baseline to 90±7 days after inclusion
  respiratory movement amplitude assessed by respiratory rate abdominal and thoracic sensors (units)
Change in psychophysiological state: alpha-rhythm index assessed by biofeedback method - from baseline to 14 days after treatment initiation | from baseline to 14 days after treatment initiation
  alpha rhythm index (%) assessed by electroencephalogram
Change in psychophysiological state: beta-rhythm index assessed by biofeedback method - from baseline to 14 days after treatment initiation | from baseline to 14 days after treatment initiation
  beta rhythm index (%) assessed by electroencephalogram
Change in psychophysiological state: alpha-rhythm index assessed by biofeedback method - from baseline to 90 days after inclusion | from baseline to 90±7 days after inclusion
  alpha rhythm index (%) assessed by electroencephalogram
Change in psychophysiological state: beta-rhythm index assessed by biofeedback method - from baseline to 90 days after inclusion | from baseline to 90±7 days after inclusion
  beta rhythm index (%) assessed by electroencephalogram
Number of participants with treatment-related adverse events assessed according to the protocol-specified adverse effects | 14 days after treatment initiation
  Number of participants with treatment-related adverse events assessed according to the Toronto Side Effects Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmila Korostovtseva, Principal Investigator — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korostovtseva L. Ischemic Stroke and Sleep: The Linking Genetic Factors. Cardiol Ther. 2021 Dec;10(2):349-375. doi: 10.1007/s40119-021-00231-9. Epub 2021 Jun 30. PMID 34191267
- [Background] Bochkarev MV, Korostovtseva LS, Medvedeva EA, Rotar OP, Sviryaev YV, Zhernakova YV, Shalnova SA, Konradi AO, Chazova IE, Boitsov SA, Shlyakhto EV. [Sleep disorders and stroke: data of the esse-rf study]. Zh Nevrol Psikhiatr Im S S Korsakova. 2019;119(4. Vyp. 2):73-80. doi: 10.17116/jnevro201911904273. Russian. PMID 31317919